CLINICAL TRIAL: NCT00762645
Title: A Twelve-Week, Double Masked, Parallel Group, Primary-Therapy Pilot Study of the Safety and Efficacy of Travoprost 0.004% Compared to Pilocarpine 1% in Patients With Chronic Angle-Closure Glaucoma
Brief Title: Travoprost 0.004% Versus Pilocarpine 1% in Patients With Chronic Angle Closure Glaucoma (CACG)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CM-06-04
Record Dates: First submitted 2008-09-24; First posted 2008-09-30 (Estimated); Results first posted 2010-03-15 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2010-03

CONDITIONS: Angle-closure Glaucoma
Keywords: IOP lowering efficacy; CACG
MeSH Terms: conditions — Glaucoma, Angle-Closure | interventions — Travoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Travoprost 0.004% (Travatan) (Experimental): One drop in each eye, once daily at 9 AM
  Interventions: Drug: Travoprost 0.004% (Travatan)
- Pilocarpine 1% (Active Comparator): One drop in each eye, forth times daily at 7 AM, 11 AM , 4 PM and 9 PM for twelve (12) weeks
  Interventions: Drug: Pilocarpine 1%

INTERVENTIONS:
Drug: Travoprost 0.004% (Travatan) — One drop in each eye, once daily at 9 AM
  Arms: Travoprost 0.004% (Travatan)
Drug: Pilocarpine 1% — One drop in each eye, forth times daily at 7 AM, 11 AM , 4 PM and 9 PM for twelve (12) weeks
  Arms: Pilocarpine 1%

SUMMARY:
The purpose of this study is to demonstrate that the Intraocular Pressure (IOP) lowering efficacy of Travoprost Ophthalmic Solution 0.004% is superior to that of Pilocarpine 1% in patients with chronic angle-closure glaucoma (CACG).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Chronic Angle Closure Glaucoma (CACG)
* 21-35 millimeters mercury mean intraocular pressure on Eligibility visit day at 9 AM
* Peripheral iridotomy performed ≥ 1 Month prior to the Screening visit
* Anterior chamber angle in which the trabecular meshwork is not visible for ≥180 degrees in gonioscopy without indentation
* Peripheral anterior synechiae (PAS)

Exclusion Criteria:

* Traumatic damage of the anterior chamber angle
* History of ocular inflammation or surgery (except for iridotomy) ≤ 3 months
* Patients who cannot be safely discontinued from use of all ocular hypotensive medication(s) for 12 days to 14 weeks
* Visual Acuity ≥ 1.0
* Contact lenses wearer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 patients were enrolled in this study
Pre-assignment Details: Patients randomized at 1:1 ratio into two treatment groups
Groups:
- Travoprost 0.004% (Travatan): Travoprost 0.004% Ophthalmic Solution
- Pilocarpine 1%: Pilocarpine 1% Ophthalmic Solution
Period: Overall Study
Arm/Group | Travoprost 0.004% (Travatan) | Pilocarpine 1%
Started | 16 | 14
Completed | 12 | 12
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Travoprost 0.004% (Travatan) | Pilocarpine 1% | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 14 | 11 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Mean Intraocular Pressure (IOP)
Time Frame: 4PM at Week 12 Visit
Measure: Mean (Standard Deviation); unit: millimeters mercury (mm Hg)
Arm/Group | Travoprost 0.004% (Travatan) | Pilocarpine 1%
Number analyzed (Participants) | 16 | 14
millimeters mercury (mm Hg) | 15.77 (2.32) | 18.35 (3.72)

2. Secondary Outcome: Number of Patients With Peripheral Anterior Synechiae (PAS)
Time Frame: Week 12 Visit
Measure: Number; unit: Participants
Arm/Group | Travoprost 0.004% (Travatan) | Pilocarpine 1%
Number analyzed (Participants) | 16 | 14
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Travoprost 0.004% (Travatan) | Pilocarpine 1%
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No